CLINICAL TRIAL: NCT03980509
Title: A "Window Trial" on Curcumin, the Active Compound in Turmeric, for Invasive Breast Cancer Primary Tumors
Brief Title: A "Window Trial" on Curcumin for Invasive Breast Cancer Primary Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103089
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Curcumin (Experimental): Curcumin will be given at 500mg by mouth twice a day, immediately after each meal. Curcumin will be given from the time surgical resection is scheduled until the night before surgical resection.
  Interventions: Drug: Curcumin

INTERVENTIONS:
Drug: Curcumin — Curcumin is an extract from turmeric

SUMMARY:
The purpose of this study is to determine whether oral administration of curcumin causes biological changes in primary tumors of breast cancer patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether oral administration of Curcuma longa extract causes biological changes related to apoptosis (DNA fragmentation) and cell proliferation (Ki67) in primary tumors of breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive breast cancer (stages I, II, or III) with primary tumor(s) ≥ 1.0 cm on mammogram, ultrasound, MRI, or physical exam
2. 18 years of age or older
3. Subject must understand risks and benefits of the protocol and be able to give informed consent
4. Women of childbearing potential (WOCBP) must agree to use an approved form of birth control and to have a negative pregnancy test result within 14 days of registration. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 consecutive months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes

   Approved forms of birth control:
   * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intra-vaginal, or transdermal)
   * progestogen only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable)
   * intrauterine device, intrauterine hormone-releasing system
   * bilateral tubal occlusion/ligation
   * vasectomized partner
   * barrier contraception
   * sexual abstinence
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Adequate hematologic and end organ function
7. Ability and capacity to comply with the study and follow-up procedures
8. Subjects must be scheduled for surgery at MUSC no less than 5 days from the planned start of day 1 and no more than 56 days from the planned start of day 1
9. At least 6 sections of unstained slides should be obtained. If sufficient slides or tissue is unavailable, the patient will be excluded from the trial

Exclusion Criteria:

1. Subjects undergoing neoadjuvant chemotherapy or neoadjuvant endocrine therapy
2. Subjects with end-stage kidney disease and/or grade II liver dysfunction
3. Subjects who are pregnant or are lactating.
4. Subjects with bile duct obstruction, gallstones, predisposition to kidney stones(39), or gastrointestinal disorders such as stomach ulcers and hyperacidity disorders(40)
5. Subjects taking anti-coagulants or platelet inhibitors
6. Subjects taking drugs metabolized by CYP3A4, CYP1A2, and CYP2A6 enzymes
7. Subjects taking drugs that interact with P-glycoprotein (P-gp)
8. Subjects taking any of the medications listed under Other Herb-Drug interactions according to the Memorial Sloan Kettering Cancer Center in section 5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Change in tumor proliferation rate | Up to 56 days
  Change in tumor proliferation rate will be based on apoptosis (DNA fragmentation) and cell proliferation (Ki67) assays in biopsies pre and post treatment with curcumin

SECONDARY OUTCOMES:
Number of adverse events reported | up to 84 days
  Safety data will be tabulated by type and grade of adverse event and will use CTCAE v. 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Nancy DeMore, MD, FACS, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No